CLINICAL TRIAL: NCT06498895
Title: Lung Ultrasound Score as Post Operative Predictive Value of Pulmonary Complications in Living Liver Transplant Recipient
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MD102/2024
Record Dates: First submitted 2024-07-06; First posted 2024-07-12 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-09

CONDITIONS: Pulmonary Complication; Post Operative Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- post operative living liver transplant recipient: lung ultrasound score will be done in first 24 hours in intensive care unit for living liver transplant recipient patient
  Interventions: Radiation: lung ultrasound

INTERVENTIONS:
Radiation: lung ultrasound — Lung ultrasound score will be done within one hour of admission,12 hours post admission then 24 hours in intensive care unit,follow up of patients will continue for 72 hours .
  a complete lung ultrasound evaluation will be performed using low frequency curved probe (2MHz-5MHz) according to the lung ultrasound score . The external lung fields will be examined by longitudinal and transverse plane scans, dividing the surface of the thorax into 12 zones: 6 on the right (anterior: upper R1 and lower R2; lateral; upper R3 and lower R4; posterior: upper R5 and lower R6) and 6 on the left side (front: upper L1 and lower L2; lateral: upper L3 and lower L4; rear: upper L5 and lower L6). LUS assigns 0 points to A lines or < 2 separate B lines plus regular sliding; 1 point with lines B ≥ 3 or spaced focal points plus regular sliding; 2 points with coalescing B lines, and 3 points to pulmonary consolidations for each zone with a score ranging from 0 (normal lungs) to 36 (worst case scenario)

SUMMARY:
The aim of this study is to determine if lung ultrasound score has a strong predictive value for post operative pulmonary complications in living liver transplant recipient

DETAILED DESCRIPTION:
Back ground :Traditional diagnostic tools such as auscultation or chest x-ray have inferior diagnostic accuracy compared to the gold standard (chest computed tomography), Lung ultrasound is becoming popular in intensive and perioperative care and there is a growing interest to evaluate its role in the detection of postoperative pulmonary pathologies.

METHODOLOGY Type of Study: observational prospective study

* Study Setting: After obtaining approval from the Research Ethical Committee of Ain Shams University, this study will be conducted in specialized Ain Shams University Hospitals.
* Study Population : living liver transplant recipient patients post operative in intensive care unit ( 25 patients ), all patients included in this study will be subjected to lung ultrasound score at the pre mentioned times (0,12,24) by most senior expert staff then follow up of patients in Intensive care unit,will reveal that patients will be divided into two groups according to occurance of lung complications to Pulmonary complications positive ( group that developed pulmonary complications ) and pulmonary complications negative (group that didn't develop pulmonary complications ) then sensitivity, specificity and predictive value of lung ultrasound score will be determined .

ELIGIBILITY:
Inclusion Criteria:

* living liver transplant recipient patients post operative in intensive care unit in first day
* Age ( Adults 21-60 )
* Sex ( both genders will be included )
* ASA 4 liver failure patients .

Exclusion Criteria:

* Presence of preoperative chronic lung diseases

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: • Study Population: living liver transplant recipient patients post operative in intensive care unit ( 25 patients ), all patients included in this study will be subjected to lung ultrasound score at the pre mentioned times (0,12,24) by most senior expert staff then follow up of patients in intensive care unit will reveal that patients will be divided into two groups according to occurance of lung complications to post operative pulmonary complications positive ( group that developed pulmonary complications ) and post operative pulmonary complications negative (group that didn't develop pulmonary complications ) then sensitivity, specificity and predictive value of lung ultrasound score will be determined
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
lung ultrasound score | first 24 hours